CLINICAL TRIAL: NCT01032135
Title: Adaptive Treatment for Alcohol and Cocaine Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807092; IND: 101,486; NCT02689674 (obsolete NCT alias)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing; Cognitive Behavioral Therapy; Counseling; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1-MI-IOP Engaged (Active Comparator): Randomized to treatment as usual, and they attend regularly but dropped out of treatment after randomization.
  Interventions: Behavioral: Motivational Interviewing
- 2-MI-IOP Non-Engaged (Experimental): Randomized to treatment as usual, and do not attend.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Telephone counseling; Behavioral: Cognitive Behavioral Therapy (CBT) Counseling; Drug: medication management; Behavioral: Intensive OutPatient Therapy
- 3-MI-PC Engaged (Active Comparator): Randomized to treatment choice, but remain attending treatment as usual then dropped out of treatment after randomization.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Telephone counseling; Behavioral: Cognitive Behavioral Therapy (CBT) Counseling
- 4-MI-PC Non-engaged (Experimental): Randomized to treatment choice, and do not attend treatment as usual, so the choice option is used.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Telephone counseling; Behavioral: Cognitive Behavioral Therapy (CBT) Counseling; Drug: medication management; Behavioral: Intensive OutPatient Therapy

INTERVENTIONS:
Behavioral: Motivational Interviewing — 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
  Other Names: MI
Behavioral: Telephone counseling — one telephone counseling session per week for 10 weeks.
  Other Names: Telephone based stepped care.
  Arms: 2-MI-IOP Non-Engaged; 3-MI-PC Engaged; 4-MI-PC Non-engaged
Behavioral: Cognitive Behavioral Therapy (CBT) Counseling — One CBT session per week, for 10 weeks.
  Other Names: CBT
  Arms: 2-MI-IOP Non-Engaged; 3-MI-PC Engaged; 4-MI-PC Non-engaged
Drug: medication management — Prescription for naltrexone
  Other Names: MM
  Arms: 2-MI-IOP Non-Engaged; 4-MI-PC Non-engaged
Behavioral: Intensive OutPatient Therapy — Return to IOP, group therapy 3 times weekly for about three hours a day.
  Other Names: IOP
  Arms: 2-MI-IOP Non-Engaged; 4-MI-PC Non-engaged

SUMMARY:
1. Primary objective #1: Determine the relative effectiveness of MI-IOP and MI-PC in the full study sample with regard to treatment engagement over weeks 1-12 and cocaine/alcohol use over weeks 1-24.

   * Hypothesis 1: An intervention that explores several possible treatment options with the patient and provides the chosen option (e.g., MI-PC) will produce higher rates of treatment engagement than an intervention focused on engagement in IOP only (e.g., MI-IOP).
   * Hypothesis 2: An intervention that explores several possible treatment options with the patient and provides the chosen option (e.g., MI-PC) will produce better cocaine/alcohol use outcomes than an intervention focused on engagement in IOP only (MI-IOP).
   * Secondary analysis 1: Among the Non-engaged patients, determine rates of selection of each of the three options in MI-PC, retention rates within each option, and cocaine/alcohol use outcomes in each option.
   * Secondary analysis 2: Among the Engaged patients, determine rates of selection of each of the three options in MI-PC, retention rates within each option, and cocaine/alcohol use outcomes in each option.
2. Primary objective #2: Determine whether the relative effectiveness of MI-IOP and MI-PC varies as a function of engagement group, with regard to treatment engagement over weeks 1-12 and cocaine/alcohol use outcomes over weeks 1-24.

   * Hypothesis 1: The predicted main effect on retention favoring MI-PC over MI-IOP will be significantly larger among patients in the Non-engaged group than among those in the Engaged group.
   * Hypothesis 2: The predicted main effect on cocaine/alcohol use outcomes favoring MI-PC over MI-IOP will be significantly larger among patients in the Non-engaged group than among those in the Engaged group.

DETAILED DESCRIPTION:
3. Secondary objective #1: Examine outcomes on three secondary measures: percent days abstinent from all substances, negative consequences of drug use, and HIV high risk behaviors.

* Hypothesis 1: Outcomes on the secondary measures will be better in MI-PC than in MI-IOP.

  4. Secondary objective #2: Test hypotheses concerning potential mediators of the predicted main effect favoring MI-PC over MI-IOP.
* Hypothesis 1: The predicted advantage of MI-PC over MI-IOP will be mediated by greater increases in motivation, self-efficacy, commitment to abstinence, and self-help involvement in MI-PC.

  5. Secondary objective #3: Test hypotheses concerning effect of additional MI intervention after initial non-engagement persists through 12 weeks.
* Hypothesis 1: A second telephone MI intervention will produce higher rates of subsequent engagement and less cocaine use than no further MI.

ELIGIBILITY:
Inclusion Criteria:

1. meet DSM-IV criteria for lifetime cocaine or alcohol dependence and have used cocaine or alcohol in the prior 6 months;
2. be > 18 years of age;
3. be judged clinically appropriate for IOP (e.g., no current psychotic disorder or evidence of severe dementia, and no acute medical problem requiring inpatient treatment;
4. have no regular IV heroin use during the past year;
5. have access to a telephone;
6. be willing to be randomized and participate in research; and
7. no current participation in methadone or other forms of DA treatment, other than IOP. Finally, because of study follow-up requirements, subjects will
8. be required to be metropolitan area residents, and
9. be able to provide the name, verified telephone number, and address of at least two contacts who can provide locator information on the patient during follow-up. We will include patients with dependence on other substances, provided that they are cocaine dependent and meet other inclusion criteria.

Exclusion Criteria:

1. have a current psychotic disorder (as assessed with the psychotic screen from the MINI) or evidence of dementia severe enough to prevent participation in outpatient treatment;
2. have acute medical problem requiring immediate inpatient treatment; or
3. are currently participating in methadone or other forms of DA treatment, other than IOP.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. McKay, Ph.D, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - VAMC, Philadelphia, Pennsylvania
  - NorthEast Treatment Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were enrolled when they entered IOP treatment. We collected baseline measures and monitored their treatment attendance. At 2 weeks, we determined whether they were engaged or nonengaged and randomized all participants at that time. Only those that were nonengaged at week 2 and still nonengaged at week 8 were rerandomized at week 8.
Groups:
- Engaged: Engaged at week 2 and remained engaged throughout the 8 weeks of study participation.
  This group did not receive any treatment intervention.
- MI-PC Non-engaged at 2 Weeks: Participants start at IOP, but at 2 weeks are not engaged. Randomized to treatment choice:
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  Medication management: Prescription for naltrexone
  Intensive OutPatient Therapy: Return to IOP, group therapy 3 times weekly for about three hours a day.
- MI-IOP Non-Engaged at 2 Weeks: Participants begin at IOP, but at 2 weeks are determined to no longer be engaged.
  Randomized to IOP
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
- MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks: Randomized to treatment choice, but remain attending treatment as usual then dropped out of treatment after randomization.
  Motivational Interviewing: 2 sessions at time of disengagement presenting treatment choices to participants.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  Medication Management: Prescription for Naltrexone
- MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks: Initially engaged at IOP, but become nonengaged in weeks 3 - 8.
  Motivational Interviewing: 2 sessions at time of disengagement.
  Return to IOP therapy 3 times weekly for three hours a day
- MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks: Began study in IOP but was nonengaged at week 2. Randomized to Patient Choice.
  Motivational Interviewing: 2 sessions at week 2 presenting treatment choices to participants.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  Medication Management: Prescription for Naltrexone
- No Further Intervention: Not engaged at week 2 and still not engaged at week 8.
  Randomized to receive no further study intervention.
Period: 2 Week Randomization
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Started | 311 | 93 | 96 | 0 | 0 | 0 | 0
Completed | 311 | 93 | 96 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 8 Week Randomization
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Started | 227 | 0 | 0 | 41 | 43 | 48 | 54
12 Week Follow up | 217 (These participants were'nt included in analyses as they didn't meet criteria for study intervention.) | 0 | 0 | 34 | 38 | 36 | 41
Completed | 201 (These participants were'nt included in analyses as they didn't meet criteria for study intervention.) | 0 | 0 | 30 | 34 | 31 | 36
Not Completed | 26 | 0 | 0 | 11 | 9 | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Engaged: Participants began treatment in IOP, consistently remained engaged in IOP throughout the study time period. This group did not reach the threshold of needing study intervention.
- MI-PC Non-Engaged: Participants began treatment in IOP but were not engaged at week 2. Randomized to receive patient choice.
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  medication management: Prescription for naltrexone
  Intensive OutPatient Therapy: Return to IOP, group therapy 3 times weekly for about three hours a day.
- MI-IOP Non-Engaged: Participants began treatment in IOP but were not engaged at week 2. Randomized back to IOP.
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
- MI-PC Engaged at 2 Weeks, Non-engaged Before 8 Weeks: Participants began treatment in IOP and were engaged at week 2. However, they dropped out of treatment between weeks 3 - 8. Randomized to Patient Choice.
  Motivational Interviewing: 2 sessions at week 2.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  medication management: Prescription for naltrexone
  Intensive OutPatient Therapy: Return to IOP, group therapy 3 times weekly for about three hours a day.
- MI-IOP Engaged at 2 Weeks, Non-engaged Before 8 Weeks: Participants began treatment in IOP and were engaged at week 2. However, they dropped out of treatment between weeks 3 - 8. Randomized back to IOP.
  Motivational Interviewing: 2 sessions at week 2.
- Total: Total of all reporting groups
Arm/Group | Engaged | MI-PC Non-Engaged | MI-IOP Non-Engaged | MI-PC Engaged at 2 Weeks, Non-engaged Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Non-engaged Before 8 Weeks | Total
Number analyzed (Participants) | 227 | 93 | 96 | 41 | 43 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 224 | 91 | 94 | 41 | 43 | 493
  >=65 years | 3 | 2 | 2 | 0 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (8.35) | 48.02 (9.84) | 47.7 (9.38) | 47.8 (9.42) | 48.5 (9.64) | 48.29 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 21 | 21 | 8 | 9 | 95
  Male | 191 | 72 | 75 | 33 | 34 | 405
Region of Enrollment [Number; unit: participants]
  United States | 227 | 93 | 96 | 41 | 43 | 500

OUTCOME MEASURES:

1. Primary Outcome: Treatment Engagement
Description: Number of treatment sessions attended
Time Frame: weeks 3 - 12
Measure: Mean (Standard Deviation); unit: treatment days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 93 | 96 | 0 | 0 | 0 | 0
treatment days |  | 3.92 (3.27) | 3.50 (3.23) |  |  |  |
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; Test type: Other; p = 0.11, Chi-squared

2. Primary Outcome: Treatment Engagement for Participants Engaged at 2 Weeks, But Disengage Before 8 Weeks
Description: Number of treatment sessions attended
Time Frame: weeks 9 - 12
Measure: Mean (Standard Deviation); unit: treatment days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 34 | 38 | 0 | 0
treatment days |  |  |  | 1.28 (1.55) | 0.76 (1.25) |  |
Statistical Analysis 1: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; Test type: Other; p = 0.02, Chi-squared

3. Primary Outcome: Treatment Engagement of Those Non-engaged at 2 Weeks and at 8 Weeks
Description: Number of treatment sessions attended
Time Frame: weeks 9 - 12
Measure: Mean (Standard Deviation); unit: treatment days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 36 | 41
treatment days |  |  |  |  |  | 0.58 (1.11) | 0.30 (0.76)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; Test type: Other; p = 0.005, Chi-squared

4. Primary Outcome: Any Drinking Days in Previous Month
Description: Days of any drinking in previous month, as reported on Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample drank in the follow up period.
Time Frame: Month 2 (weeks 5 - 8 post baseline)
Population: The number of participants analyzed represents the number that were available to provide research data. Those participants who were engaged and remained engaged in treatment were not included in these analyses.
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 70 | 63 | 28 | 37 | 30 | 32
proportion of participants |  | 0.57 (0.50) | 0.37 (0.49) | 0.46 (0.51) | 0.41 (0.50) | 0.60 (0.50) | 0.63 (0.49)

5. Primary Outcome: Any Drinking Days in Previous Month
Description: Any drinking days during previous month, as reported on Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample drank in the follow up period.
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 72 | 62 | 28 | 36 | 29 | 34
proportion of participants |  | 0.58 (0.50) | 0.37 (0.49) | 0.57 (0.50) | 0.42 (0.50) | 0.72 (0.45) | 0.50 (0.51)

6. Primary Outcome: Any Drinking
Description: Any drinking at follow up, as reported on Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample drank in the follow up period.
Time Frame: Month 4 (weeks 13 - 15 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.49 (0.50) | 0.26 (0.44) | 0.42 (0.50) | 0.30 (0.47) | 0.50 (0.51) | 0.47 (0.51)

7. Primary Outcome: Any Drinking
Description: Any drinking at follow up, as reported on Time Line Follow Back, This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample drank in the follow up period.
Time Frame: Month 5 (weeks 16 - 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.51 (0.50) | 0.31 (0.47) | 0.42 (0.50) | 0.30 (0.47) | 0.42 (0.50) | 0.57 (0.50)

8. Primary Outcome: Any Drinking
Description: as for outcome 6
Time Frame: Month 6 (weeks 21 - 24 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.56 (0.50) | 0.31 (0.47) | 0.50 (0.51) | 0.27 (0.45) | 0.42 (0.50) | 0.63 (0.49)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.0007, Chi-squared; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.23 to 0.68]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.16, Chi-squared; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.23 to 1.27]
Statistical Analysis 3: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.79, Chi-squared; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.48 to 2.60]

9. Primary Outcome: Percent Days Drinking
Description: Percent days of any drinking at follow up, from Time Line Follow Back
Time Frame: Month 2 (weeks 5 - 8 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 70 | 63 | 28 | 37 | 30 | 32
percentage of days |  | 12.81 (18.10) | 12.93 (26.81) | 17.35 (29.12) | 8.11 (15.12) | 20.00 (28.15) | 17.30 (25.80)

10. Primary Outcome: Percent Days Drinking
Description: Percent days of any drinking at follow up, from Time Line Follow Back
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 72 | 62 | 28 | 36 | 29 | 34
percentage of days |  | 14.51 (26.89) | 9.10 (21.68) | 15.31 (25.49) | 8.23 (15.24) | 20.02 (29.61) | 11.66 (23.50)

11. Primary Outcome: Percent Days Drinking
Description: Percent days of any drinking at follow up, from Time Line Follow Back
Time Frame: Month 4 (weeks 13 - 16 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 15.76 (26.16) | 8.96 (24.65) | 21.13 (37.69) | 13.42 (29.38) | 6.37 (11.55) | 18.81 (31.37)

12. Primary Outcome: Percent Days Drinking
Description: Percent days of any drinking at follow up, fromTime Line Follow Back
Time Frame: Month 5 (weeks 17 - 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 18.37 (29.86) | 8.22 (19.78) | 20.24 (33.31) | 11.47 (28.57) | 6.99 (15.09) | 20.60 (27.90)

13. Primary Outcome: Percent Days Drinking
Description: Percent days of any drinking at follow up, from Time Line Follow Back
Time Frame: Month 6 (weeks 21 - 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 14.75 (26.05) | 5.66 (16.61) | 19.05 (34.19) | 8.77 (24.42) | 8.70 (21.67) | 15.38 (23.06)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.009, Chi-squared; Odds Ratio (OR) = -1.08, 95% CI 2-sided [-1.87 to -0.29]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.23, Chi-squared; Odds Ratio (OR) = -0.84, 95% CI 2-sided [-2.20 to 0.52]
Statistical Analysis 3: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.58, Chi-squared; Odds Ratio (OR) = -0.34, 95% CI 2-sided [-1.52 to 0.85]

14. Primary Outcome: Any Heavy Drinking Days
Description: days of five or more drinks per drinking day for men, four or more drinks per drinking day for women, at follow up, from Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of heavy drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample engaged in heavy drinking in the follow up period.
Time Frame: Month 2 (weeks 5 - 8 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 70 | 63 | 28 | 37 | 30 | 32
proportion of participants |  | 0.49 (0.50) | 0.24 (0.43) | 0.36 (0.49) | 0.24 (0.43) | 0.47 (0.51) | 0.34 (0.48)

15. Primary Outcome: Any Heavy Drinking Days
Description: five or more drinks per drinking day for men, four or more drinks per drinking day for women, at follow up, from Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of heavy drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample engaged in heavy drinking in the follow up period.
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 72 | 62 | 28 | 36 | 29 | 34
proportion of participants |  | 0.44 (0.50) | 0.26 (0.44) | 0.36 (0.49) | 0.33 (0.48) | 0.55 (0.51) | 0.32 (0.47)

16. Primary Outcome: Any Heavy Drinking Days
Description: five or more drinks per drinking day for men, four or more drinks per drinking day for women at follow up, from Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of heavy drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample engaged in heavy drinking in the follow up period.
Time Frame: Month 4 (weeks 13 - 16 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.37 (0.49) | 0.15 (0.36) | 0.38 (0.49) | 0.24 (0.44) | 0.38 (0.49) | 0.27 (0.45)

17. Primary Outcome: Any Heavy Drinking Days
Description: five or more drinks per day for men, four or more drinks per day for women, from Time Line Follow Back. This is a dichotomous measure, so the means that are reported are the percentage of people who have had any days of heavy drinking during the follow up period specified. In other words, 0.57 indicates that 57% of the sample engaged in heavy drinking in the follow up period.
Time Frame: Month 5 (weeks 17 to 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.37 (0.49) | 0.19 (0.39) | 0.38 (0.49) | 0.24 (0.44) | 0.25 (0.44) | 0.33 (0.48)

18. Primary Outcome: Any Heavy Drinking Days
Description: as for outcome 17
Time Frame: Month 6 (weeks 21 - 24 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 54 | 24 | 33 | 24 | 30
proportion of participants |  | 0.43 (0.50) | 0.17 (0.38) | 0.38 (0.49) | 0.21 (0.42) | 0.25 (0.44) | 0.37 (0.49)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.0001, Chi-squared; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.19 to 0.58]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.36, Chi-squared; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.29 to 1.54]
Statistical Analysis 3: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.45, Chi-squared; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.58 to 3.54]

19. Primary Outcome: Percent Days Heavy Drinking
Description: Percent days heavy drinking at follow up, from Time Line Follow Back
  *heavy drinking is defined as five or more drinks per day for men, four or more for women
Time Frame: Month 2 (weeks 5 - 8 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 70 | 63 | 28 | 37 | 30 | 32
percentage of days |  | 11.73 (18.28) | 7.14 (20.11) | 10.59 (22.13) | 6.37 (14.85) | 12.98 (22.48) | 10.49 (21.16)

20. Primary Outcome: Percent Days Heavy Drinking
Description: Percent days heavy drinking at follow up, from Time Line Follow Back
  * heavy drinking is defined as five or more drinks per day for men, four or more for women.
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 72 | 62 | 28 | 36 | 29 | 34
percentage of days |  | 10.58 (22.61) | 6.05 (17.92) | 12.37 (24.33) | 5.65 (14.09) | 14.16 (24.53) | 3.99 (9.04)

21. Primary Outcome: Percent Days Heavy Drinking
Description: Percent days heavy drinking at follow up, from Time Line Follow Back
  *heavy drinking is defined as five or more drinks per drinking day for men, four or more for women
Time Frame: Month 4 (weeks 13 - 16 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 11.56 (23.55) | 7.01 (23.15) | 20.98 (37.77) | 8.98 (24.84) | 5.75 (11.73) | 13.93 (30.18)

22. Primary Outcome: Percent Days Heavy Drinking
Description: Percent days heavy drinking at follow up, from Time Line Follow Back
  * heavy drinking is defined as five or more drinks per drinking day for men, four or more for women
Time Frame: Month 5 ( weeks 17 - 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 13.49 (27.37) | 5.73 (18.48) | 20.09 (33.40) | 8.33 (24.48) | 5.43 (15.19) | 15.12 (28.18)

23. Primary Outcome: Percent Days Heavy Drinking
Description: as for outcome 21
Time Frame: Month 6 (weeks 21 - 24 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 63 | 53 | 24 | 33 | 23 | 30
percentage of days |  | 11.30 (23.91) | 3.77 (15.34) | 18.3 (34.52) | 5.74 (19.25) | 7.61 (21.73) | 10.87 (22.86)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.003, Chi-squared; Odds Ratio (OR) = -1.09, 95% CI 2-sided [-1.80 to -0.39]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.10, Chi-squared; Odds Ratio (OR) = 0.02, 95% CI 2-sided [-1.10 to 1.14]

24. Primary Outcome: Any Cocaine Use
Description: Any cocaine using self report, binary measure of percent days cocaine use.
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 83 | 76 | 26 | 33 | 29 | 35
proportion of participants |  | 0.45 (0.50) | 0.42 (0.50) | 0.31 (0.47) | 0.36 (0.49) | 0.66 (0.48) | 0.46 (0.51)

25. Primary Outcome: Any Cocaine Use
Description: Any cocaine using self report, binary measure of percent days cocaine use
Time Frame: Month 4 (weeks 13 - 16 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 65 | 51 | 23 | 30 | 24 | 31
proportion of participants |  | 0.43 (0.50) | 0.29 (0.46) | 0.39 (0.50) | 0.23 (0.43) | 0.63 (0.49) | 0.45 (0.51)

26. Primary Outcome: Any Cocaine Use
Description: Any cocaine using self report, binary measure of percent days cocaine use
Time Frame: Month 5 (weeks 17 - 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 65 | 52 | 23 | 30 | 24 | 31
proportion of participants |  | 0.45 (0.50) | 0.35 (0.48) | 0.35 (0.49) | 0.23 (0.43) | 0.58 (0.50) | 0.42 (0.50)

27. Primary Outcome: Any Cocaine Use
Description: Any cocaine using self report, binary measure of percent days cocaine use
Time Frame: Month 6 (weeks 21 - 24 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 52 | 65 | 23 | 30 | 24 | 31
proportion of participants |  | 0.35 (0.48) | 0.49 (0.50) | 0.35 (0.49) | 0.30 (0.47) | 0.54 (0.51) | 0.58 (0.50)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.13, Chi-squared; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.38 to 1.14]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.71, Chi-squared; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.33 to 2.12]
Statistical Analysis 3: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.36, Chi-squared; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.64 to 3.40]

28. Primary Outcome: Percent Days Cocaine Use
Description: Percent days of any cocaine use, self reported
Time Frame: Month 3 (weeks 9 - 12 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 74 | 60 | 26 | 33 | 30 | 35
percentage of days |  | 12.61 (25.38) | 9.35 (20.19) | 11.68 (25.33) | 3.90 (7.54) | 18.45 (28.68) | 12.35 (23.39)

29. Primary Outcome: Percent Days Cocaine Use
Description: Percent days of any cocaine use, self reported
Time Frame: Month 5 (weeks 17 - 20 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 68 | 53 | 23 | 31 | 25 | 33
percentage of days |  | 10.87 (23.78) | 12.60 (28.40) | 14.60 (27.00) | 4.26 (17.99) | 19.14 (33.07) | 15.26 (28.28)

30. Primary Outcome: Percent Days Cocaine Use
Description: Percent days of any cocaine use, self reported
Time Frame: Month 6 (weeks 21 - 24 post baseline)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks | No Further Intervention
Number analyzed (Participants) | 0 | 68 | 53 | 23 | 31 | 25 | 33
percentage of days |  | 7.76 (16.00) | 9.50 (24.27) | 10.09 (22.40) | 4.95 (13.19) | 15.57 (28.02) | 13.35 (26.10)
Statistical Analysis 1: Comparison: MI-PC Non-engaged at 2 Weeks vs MI-IOP Non-Engaged at 2 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.75, Chi-squared; Odds Ratio (OR) = -0.13, 95% CI 2-sided [-0.94 to 0.60]
Statistical Analysis 2: Comparison: MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks vs MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.16, Chi-squared; Odds Ratio (OR) = -0.84, 95% CI 2-sided [-1.98 to 0.30]
Statistical Analysis 3: Comparison: MI-PC Non-engaged at 2 Weeks, Still Non-engaged at 8 Weeks vs No Further Intervention; The statistical analyses used data from all follow up assessments; Test type: Other; p = 0.42, Chi-squared; Odds Ratio (OR) = 0.60, 95% CI 2-sided [-0.85 to 2.04]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- MI-PC Non-engaged at 2 Weeks: Participants start at IOP, but at 2 weeks are non-engaged.
  Randomized to treatment choice:
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  Medication Management: Prescription for naltrexone
  Intensive OutPatient Therapy: Return to IOP, group therapy 3 times weekly for about three hours a day.
- MI-IOP Non-Engaged at 2 Weeks: Participants start at IOP, but at 2 weeks are non-engaged.
  Randomized to IOP
  Motivational Interviewing: 2 sessions at week 2, potential 2 sessions at week 8 if the participant drops out.
- MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks: Participants start at IOP, Engaged at 2 weeks but disengage between 3 - 8 weeks.
  Randomized to treatment choice:
  Motivational Interviewing: 2 sessions at week 2
  Telephone counseling: one telephone counseling session per week for 10 weeks.
  Cognitive Behavioral Therapy (CBT) Counseling: One CBT session per week, for 10 weeks.
  Medication Management: Prescription for naltrexone
  Intensive OutPatient Therapy: Return to IOP, group therapy 3 times weekly for about three hours a day.
- MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks: Initially engaged at IOP, but become non-engaged in weeks 3 - 8.
  Randomized to IOP
  Motivational Interviewing: 2 sessions at week 2
Arm/Group | Engaged | MI-PC Non-engaged at 2 Weeks | MI-IOP Non-Engaged at 2 Weeks | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/93 | 0/96 | 1/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 34/227 | 16/93 | 9/96 | 4/41 | 4/43
Other Adverse Events (participants affected / at risk) | 0/227 | 0/93 | 0/96 | 0/41 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engaged (N=227) | MI-PC Non-engaged at 2 Weeks (N=93) | MI-IOP Non-Engaged at 2 Weeks (N=96) | MI-PC Engaged at 2 Weeks, Disengage Before 8 Weeks (N=41) | MI-IOP Engaged at 2 Weeks, Disengage Before 8 Weeks (N=43)
Hospitalizations (General disorders) | 34 | 16 | 9 | 4 | 4 — The SAEs reported ranged from suicide attempts and depression, to detox and overdose, to migraines. The SAEs were found from searches of electronic medical records and were not study related. The participants were not receiving interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No